CLINICAL TRIAL: NCT00748826
Title: Remicade Safety Line
Brief Title: Remicade Safety Line (Study P03236)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P03236
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab -Rheumatoid Arthritis Participants
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Patients with active rheumatoid arthritis (RA) confirmed with American College of Rheumatology (ACR) criteria could take part in the project if they did not respond sufficiently to disease-modifying products, including methotrexate, received Infliximab administration as intravenous (IV) infusion over a period of two hours. Dosage and infusion intervals were employed in accordance to the Summary of Product Characteristics (SmPC): 5 mg/kg body weight at week 0 of
  Infliximab therapy with additional infusions of 5 mg/kg at week 2
  Other Names: Remicade

SUMMARY:
The goal of this study is to implement instruments that would increase the treating physician's awareness of the necessary tuberculosis screening when starting a new patient on infliximab (Remicade) therapy who has not reacted sufficiently to disease-modifying preparations, including methotrexate.

DETAILED DESCRIPTION:
This study used a non-probability sampling method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active rheumatoid arthritis confirmed with adequate clinical response(ACR) criteria who did not react sufficiently to disease-modifying preparations, including methotrexate, and who are receiving new treatment with infliximab.

Exclusion Criteria:

* As per Summary of Product Characteristics (SmPC)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The goal is to document all patients in the clinic that meet the inclusion criteria within the scope of the project.
Sampling Method: Non-Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2002-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 508 rheumatoid arthritis participants initially enrolled on study. An additional 68 participants with psoriatic arthritis (PsA) were enrolled but were not included in the analyses.
Groups:
- Infliximab: Patients with active rheumatoid arthritis (RA) confirmed with ACR criteria could take part in the project if they did not respond sufficiently to disease-modifying products, including methotrexate, received Infliximab administration as intravenous (IV) infusion over a period of two hours. Dosage and infusion intervals were employed in accordance to the Summary of Product Characteristics (SmPC): 5 mg/kg body weight at week 0 of Infliximab therapy with additional infusions of 5 mg/kg at week 2
Period: Overall Study
Arm/Group | Infliximab
Started | 508 (Of 576 total enrolled, 68 out of scope participants were not used for analyses)
Completed | 207
Not Completed | 301

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 508
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.80 (13.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 357
  Male | 151

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had the Mendel Mantoux Test as the First Screening Test for Active or Latent Tuberculosis (TB) Before Starting Treatment
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). The number of participants who had the Mendel Mantoux test (Tuberculin sensitivity skin test by intradermal injection) per clinical testing as the first screening test was presented in
  three categories:
  * Yes
  * No
  * Missing
Time Frame: Baseline
Population: Of 576 participants enrolled on study (508 with rheumatoid arthritis and 68 with psoriatic arthritis), only data from the 508 rheumatoid arthritis participants was evaluated.
Measure: Number; unit: participants
Arm/Group | Infliximab
Number analyzed (Participants) | 508
participants
  Yes | 481
  No | 26
  Missing | 1

2. Primary Outcome: Number of Participants Who Had the Tine Test as the First Screening Test for Active or Latent Tuberculosis Before Starting Treatment
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). The number of participants who had the Tine test (Multiple puncture Tuberculin skin test) per clinical testing as the first screening test was presented in three categories:
  * Yes
  * No
  * Missing
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Infliximab
Number analyzed (Participants) | 508
participants
  Yes | 23
  No | 484
  Missing | 1

3. Primary Outcome: Number of Participants Who Had the In-vitro TB Test as the First Screening Test for Active or Latent Tuberculosis Before Starting Treatment
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). The number of participants who had the In-vitro TB test (cellular blood test, i.e. gamma interferon release assays) per clinical testing as the first screening test was presented in three categories:
  * Yes
  * No
  * Missing
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Infliximab
Number analyzed (Participants) | 508
participants
  Yes | 6
  No | 216
  Missing | 286

4. Primary Outcome: Number of Participants Who Had a Chest X-ray as Part of TB Screening for Active or Latent Tuberculosis Before Starting Treatment
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). If done according to guidelines, complete TB screening comprised of a TB screening test and a chest X-ray. The number of participants who had a frontal chest X-ray was presented in three categories:
  * Yes
  * No
  * Missing
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Infliximab
Number analyzed (Participants) | 508
participant
  Yes | 459
  No | 48
  Missing | 1

ADVERSE EVENTS:
Arm/Group | Infliximab
Serious Adverse Events (participants affected / at risk) | 1/508
Other Adverse Events (participants affected / at risk) | 0/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=508)
Myocardial Infarction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial results belong to the SPONSOR only, all investigators are not allowed to publish trial results without permission of the SPONSOR.